CLINICAL TRIAL: NCT03447288
Title: Incidence of Dyssynchronous Spontaneous Breathing Effort, Breath-stacking and Reverse Triggering in Early ARDS
Brief Title: Incidence of Dyssynchronies in Early ARDS
Acronym: BEARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-182
Record Dates: First submitted 2017-07-05; First posted 2018-02-27 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: ARDS; Acute Hypoxemic Respiratory Failure
Keywords: Dyssynchrony; Breath-stacking; Asynchrony; Reverse Triggering; Mechanical Ventilation; Sedation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients sedated under mechanical ventilation with acute hypoxemic respiratory failure with a PaO2/FiO2 equal or less than 200mmHg (Acute Respiratory Distress Syndrome, ARDS and non-ARDS) will be included in the study early in the course of the disease (first week of mechanical ventilation). At enrollment, data on the clinical condition of the patient will be recorded together with ventilation settings: ventilation mode, the fraction of inspired oxygen (FiO2), PEEP, tidal volume, set pressure, respiratory rate, time of the respiratory cycle, recent blood gas parameters.

Airway pressure, flow, and esophageal pressure (or alternatively electrical activity of the diaphragm, Eadi) will be recorded 3 times a day for 7 days:

1. Period 1 (morning): duration 20-30 minutes
2. Period 2 (afternoon): duration 20-30 minutes
3. Period 3 (evening / night): duration 20-30 minutes

Registration will be ended at extubation, death or at eight days from the first recording.

Monitoring of vital parameters (hemodynamic and respiratory) will be continuous throughout the duration of the study, as per normal clinical practice. All drugs used during the day of the measurements will be recorded. The patient will then be followed until discharge from the ICU and after 60 days of discharge to evaluate mortality.

As an ancillary study, in a subgroup of patients continuous simplified measurement of respiratory recordings together with hourly clinical data on sedation and extended simplified polysomnography recordings will be performed within the first 7 days from inclusion.

The analysis of the recorded waveforms will be performed in a single center by a centralized system that will quantify dyssynchrony and its intensity, calculate pressure time product, collect clinical and physiological data and outcome, and investigate possible correlations.

DETAILED DESCRIPTION:
Measurements

Physiological measurements Airway pressure, esophageal pressure, electrical activity of the diaphragm and flow

1. Flow and airway pressure signal will be recorded from the ventilators by connecting the ventilator to a laptop computer if possible. Recording these data simultaneously with esophageal pressure or electrical activity of the diaphragm (see later in protocol for details) could be technically unfeasible. In this case, a flow sensor and an additional port for pressure measurement will be connected to the endotracheal tube proximal to the Y connector (without interfering with patient's breathing). Both, flow sensor and pressure port will be connected to differential pressure transducers respectively. Signals will be acquired with at least 100 Hz sampling.
2. In centers used to perform esophageal pressure measurements, an esophageal catheter will be inserted as per usual clinical practice, checked for accuracy with an occlusion test, and connected to a 3 ways stopcock and a pressure transducer. The occlusion test will be recorded and performed before any new recordings. Any ventilator can be used if an esophageal pressure is used.
3. If available, in centers used to record or monitor the electrical activity of the diaphragm, instead of an esophageal catheter, the electrical activity of the diaphragm will be provided by a catheter dedicated to the monitoring of the electrical activity of the diaphragm, or EaDi, on a Servo-I or Servo-U ventilator (Maquet©, Lund, Sweden). This catheter is formally designed to be used for a specific mode of ventilation called Neurally Adjusted Ventilatory Assist (NAVA) but here will be used for monitoring purposes only (NAVA catheter). In such cases a specific software (Servotracker, Maquet) may be used to record all signals from the ventilator.
4. In case the patient has been enrolled but the esophageal catheter cannot be placed or is contraindicated, the recordings will be limited to airway pressure and flow. Each centre should have a minimum of 5 patients with esophageal catheter or electrical activity recording.
5. As an ancillary study, in a subgroup of patients, simplified recordings will be obtained only flow and airway pressure signals will be performed continuously directly taken from the ventilator by connecting the ventilator to a laptop computer equipped with a special software for off line analysis (Better Care ©, Sabadell, Spain).
6. Occlusion pressure (or pressure at 0.1 sec, P0.1) as an index of respiratory drive. In patients triggering the ventilator, the P0.1 will be analyzed from the tracings. The only condition to have reliable measurements is to use a pressure triggering, not a flow triggering.

As an ancillary study, in a subgroup of patients, a simplified extended polysomnography recording will be performed during the first 7 days after inclusion using a home polysomnography device (Prodigy, CerebraHealth ©, Canada) equipped with 2 frontal EEG a reference electrode to the mastoid, EMG, and electrooculogram.

Data collection

At the beginning of the recordings, ventilatory settings will be collected: ventilator brand, mode of ventilation and settings including: FiO2, PEEP, set and real tidal volume (or pressure), set and real respiratory rate, maximum inspiratory flow, inspiratory time, Glasgow coma scale and Richmond Agitation Sedation Scale (RASS) or Riker Sedation Agitation Scale (SAS). Any medications used at the day of the measurement and before will be collected especially neuromuscular blocking agents, sedatives (brands and doses), opiates and vasopressors including dose, duration of the treatment and date of last use. Investigators will also collect clinical characteristics of the patients (SAPS and SOFA at ICU admission and at the day of the recording, main ARDS or AHRF etiology and risk factors, age, gender, weight, height, days of mechanical ventilation, patient's position -supine vs prone-, kidney and liver function). Other comorbidities will be recorded, with special emphasis in the ones that could affect the incidence of the studied phenomenon, such as: COPD, lung transplant or any neuromuscular condition that could affect the respiratory drive or respiratory muscle function.

Patients will be followed up to get the total duration of mechanical ventilation, ICU length of stay, day of the first weaning attempt, day of tracheotomy if any, status at ICU discharge (alive or death) and at hospital discharge and at day 60.

ELIGIBILITY:
Inclusion Criteria:

* Moderate and severe ARDS and AHRF, according to the Berlin definition. The absence of the Chest X-Ray criterion (e.g. unilateral disease) or the presence of primary cardiac dysfunction will define AHRF.
* Continuous intravenous sedation
* Deep sedation: Richmond Agitation Sedation Scale (RASS) ≤ -3 or Riker Sedation-Agitation Scale (SAS) ≤ 3

Exclusion Criteria:

* <18 years
* Patients with a significant bronchopleural fistula
* Pure COPD exacerbation
* Patients on chronic home ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe acute hypoxemic respiratory failure (ARDS and non-ARDS) under sedation and mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dyssynchrony | Within 1 Year
  For each patients, the number of dyssynchrony (reverse triggering, breath stacking, short cycles) will be counted over the recorded period. An asynchrony index, (number of dyssynchrony divided by the total number of breaths) as well as the number of dyssynchrony per minute will be calculated globally and for each dyssynchrony type.
  Patients with ARDS will be compared to patients with AHRF. Patients with severe ARDS or severe AHRF (<120) will be compared to less severe patients.

SECONDARY OUTCOMES:
Intensity of dyssynchrony | Within 1 Year
  Assessement of the frequency and magnitude of effort assessed by esophageal pressure or electrical activity of he diaphragm for each type of dyssynchrony
Correlation of clinical outcome with intensity of dyssynchrony | Within 1 Year
  Outcomes will be the duration of mechanical ventilation (in days); the number of ventilator-free days at day 28 (number of days alive without mechanical ventilation in 28 days; death equals 0 ventilator-free days); ICU survival and hospital survival. For each type of dyssynchrony, the outcomes will be correlated with the intensity of dyssynchrony.
  Intensity of dyssynchrony will be based on the dyssynchrony index above a minimal level of effort for each dyssynchrony.
  The outcomes above several thresholds of dyssynchrony index (10%, 30%, 50%) will be compared.
Impact of reverse triggering on breathing effort | Within 1 Year
  The breathing effort (pressure-time product) will be calculated and its value will be compared for breaths with and without reverse triggering.
Quantification of spontaneous breathing efforts associated with dyssynchronies. | Within 1 Year
  For each dyssynchrony found, the effort measured by the pressure-time product using esophageal pressure will be calculated. And the clinically relevant dyssynchronies will be determined based on a minimal amount of effort.
Association between pH and Dyssynchrony | Within 1 Year
  Arterial pH will be compared at different values of dyssynchrony index above a minimal level (10%, 30% and 50%).
Association between sedation and Dyssynchrony | Within 1 Year
  Level of sedation (assessed either Sedation Agitation Score "SAS" or the Richmond Agitation and Sedation Scale "RASS") by the will be compared at different values of dyssynchrony index above a minimal level (10%, 30% and 50%).
Association between sedatives and Dyssynchrony | Within 1 Year
  Values of dyssynchrony index above a minimal level will be compared between patients receiving primarily propofol versus benzodiazepines.
Clusters of dyssynchronies | Within 1 Year
  Timing of detection of dyssynchrony
Sleep depth measured with EEG | Within 1 Year
  As part of an ancillary exploratory study, various measures of brain activity, using EEG derived parameters including distribution of sleep depth using an automated scoring system named Odds Ratio Product (ORP) will be studied. ORP score ranges from 0 (corresponding to deep sleep) to 2.5 (corresponding to full wakefulness).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, Dr., Principal Investigator — Unity Health Toronto
Locations (14):
- Canada (2):
  - St Michael's hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China
- Centre Hospitalier Universitaire - CHU Angers, Angers, France
- Universitätsklinikum Schleswig-Holstein, Kiel, Germany
- University Hospital of Heraklion, Heraklion, Greece
- Italy (4):
  - University of Ferrara, Ferrara
  - Azienda Ospedaliero - Universitaria OORR Ospedali Riuniti di Foggia, Foggia
  - ASST Santi Paolo e Carlo, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
- VU University Medical Centre Amsterdam, Amsterdam, Netherlands
- Vall d'Hebron University Hospital, Barcelona, Spain
- National Cheng-Kung University and Hospital, Tainan, Taiwan
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share physiologic tracings with no participant identification.

REFERENCES:
- [Derived] Bianchi I, Grassi A, Pham T, Telias I, Teggia Droghi M, Vieira F, Jonkman A, Brochard L, Bellani G. Reliability of plateau pressure during patient-triggered assisted ventilation. Analysis of a multicentre database. J Crit Care. 2022 Apr;68:96-103. doi: 10.1016/j.jcrc.2021.12.002. Epub 2021 Dec 21. PMID 34952477
- [Derived] Pham T, Montanya J, Telias I, Piraino T, Magrans R, Coudroy R, Damiani LF, Mellado Artigas R, Madorno M, Blanch L, Brochard L; BEARDS study investigators. Automated detection and quantification of reverse triggering effort under mechanical ventilation. Crit Care. 2021 Feb 15;25(1):60. doi: 10.1186/s13054-020-03387-3. PMID 33588912